CLINICAL TRIAL: NCT05199077
Title: A Phase IIa Study to Investigate the Efficacy and Safety Profile of GM-XANTHO in Pressure Ulcer Patients
Brief Title: A Study of GM-XANTHO in Pressure Ulcer Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xantho Biotechnology Co., LTD (Industry)
Collaborators: Virginia Contract Research Organization Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XANGMXH20210702
Record Dates: First submitted 2021-12-27; First posted 2022-01-20 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Pressure Ulcer; Diabetes Mellitus
Keywords: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: placebo group 2.5 % GM-XANTHO of cohort A 5 % GM-XANTHO of cohort B.
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- placebo group (Placebo Comparator): Topical administration of a drug-free placebo ointment daily for 28 days.
  Interventions: Drug: GM-XANTHO
- cohort A (Active Comparator): Topical administration of a 2.5 % GM-XANTHO ointment daily for 28 days.
  Interventions: Drug: GM-XANTHO
- cohort B (Active Comparator): Topical administration of a 5 % GM-XANTHO ointment daily for 28 days.
  Interventions: Drug: GM-XANTHO

INTERVENTIONS:
Drug: GM-XANTHO — a topical applied ointment
  Other Names: Placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blind, 3-arm, single-center, phase IIa, parallel study to assess the efficacy, safety, and tolerability of topically applied 2.5%, 5% GM-XANTHO plus standard of care in patients with stage II or stage III pressure ulcer.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind,three-arm, single-centered, parallel study to evaluate the efficacy and safety profiles of the topical ointment, GM-XANTHO. For placebo group and cohort A, at least 30% eligible subjects with DM will be enrolled, for cohort B, only eligible subjects with DM will be enrolled.

Patients with pressure ulcer will be instructed to apply appropriate amount of placebo ( 3.2 mg/cm 2, for placebo group) 2.5 % GM-XANTHO [3.2 mg/cm 2, for cohort A ], or 5% GM-XANTHO [3.2 mg/cm 2, for cohort B] ointment once a day for 28 days. The appropriate dressings that maintain a moist wound as a standard background intervention.

For primary endpoint, the wound completed healing rate of the target lesion will be continuously observed to evaluate the efficacy. For secondary endpoints, the efficacy profile of GM-XANTHO will be assessed by the healing time, recurrent time and recurrent rate. The baseline of each efficacy factors will be evaluated on Day 1 before dosing.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female or male inpatients including in those staying in a long-term care facility, age ≥ 20 years old.

  2. Patient who is able to understand the nature of this study and accepts to enter the study by signing written informed consent.

  3. Patient is willing to comply with protocol-stated requirements, instructions and restrictions.

  4. Patients who have at least 1 well diagnosed Stage 2 to 3 friction-injury associated PU (according to National Pressure Ulcer Advisory Panel [NPUAP] Staging Guidelines, 2019) as the index ulcer at Screening Visit and First Dosing Visit located in any of the following regions.

  5. Surface dimensions of the index PU should be ≥ 5 cm2 and ≤ 50 cm2 as measured by the greatest length and width method through using an mm-scale ruler.

  6. Patients with adequate arterial blood flow and perfusion near the site of the injury for lower extremity ulcers (e.g., the foot is warm to the touch and has palpable pulses) 7. Patients who agree discontinuation of systemic corticosteroids and systemic immune modulating agents during the study period 8. Patients who agree discontinuation of all local treatment modalities, including but not limited to topical antimicrobials, topical corticosteroid or light treatments during the study period for/on the index wound.

  9. Patients are required to stop using treatment modalities listed in Criteria #7 and #8 at least 14 days (or longer if the treatment half-life requires so; 7 half-life should have elapsed).

  10. Patient has adequate hematopoietic, hepatic function, nutrition condition and renal function as assessed by the following laboratory requirements to be conducted within 28 days prior to the first dosing:
* Hemoglobin ≥ 10 g/dL
* Total WBC ≥ 3,000 cells/μL
* Platelet ≥ 55,000 counts/μL without transfusion support
* Total bilirubin ≤ 1.5× ULN and no sign of jaundice
* ALT and AST ≤ 5× ULN and no clinical significance
* pre-albumin ≥ 11 mg/dL
* Creatinine ≤ 1.5× ULN and no clinical significance 11. If the subject has diabetes mellitus [as per American Diabetes Association guidelines (ADA guideline, 2021)], the hemoglobin A1c (HbA1c) should be≦10 % with a stable anti-diabetes regimen (monotherapy or combination therapy including oral anti-diabetes medications) for more than 12 weeks.

  12. All male patients and female patients with child-bearing potential (between puberty and 2 years after menopause) should use at least any one of the appropriate contraception methods shown below, for during and at least 4 weeks after GM-XANTHO treatment.
  1. Total abstinence [when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].
  2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
  3. Male sterilization. For female subjects on the study, the vasectomized male partner should be the sole partner for that subject.
  4. Combination of any two of the following listed methods: (d.1+d.2 or d.1+d.3, or d.2+d.3):

  d.1 Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.

  d.2 Placement of an intrauterine device (IUD) or intrauterine system (IUS). d.3 Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

Exclusion Criteria:

* 1. Surgical treatment of pressure ulcers within 30 days prior to the Screening Visit.

  2. Patients who have any concurrent skin condition that will interfere with assessment of treatment or any condition associated with a wound healing abnormality (e.g.: connective tissue disorder or immune disorder).

  3. Patients who have active infection on the PU site(s) at baseline 4. Patients who have known hypersensitivity to the study medication 5. Patients with chronic condition(s) which either is not stable or not well controlled.

  6. Patients having positive results for HBV, HCV or HIV screens 7. Patients who are pregnant or breast feeding 8. Patients carry history of malignancy of any organ system (other than cervical carcinoma in situ or localized prostate cancer) within 5 years prior to study entry.

  9. Patients had participated in investigational drug trials and took any investigational drugs within 30 days or within 5 half-life of the investigational drugs prior to the screening visit.

  10. Patients who are not suitable to participate in the trial as judged by the Investigator(s)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
percentage change | 112 days
  percentage change in ulcer area

SECONDARY OUTCOMES:
Time to complete wound closure | 112 days
  The time from the baseline to the complete healing of the target lesion
The incidence of complete wound closure of the target lesion. | 112 days
  The percentage of subjects that achieved complete wound closure from baseline at each visit.
Time to Recurrence | 112 days
  The time from when the target lesion is completely healed to a new ulcer occurred at the same location
Recurrent rate | 112 days
  The incidence of ulcer recurrence at each visit.
Changes in wound status | 112 days
  Changes in wound status by Pressure Ulcer Scale for Healing (PUSH) tool
Change in pain score of the target lesion from baseline | 112 days
  Change in pain score of the target lesion from baseline by using the Visual Analog Scale (VAS)
The Quality of Life | 112 days
  The Quality of Life by using the Short Form (SF)-36 Health Survey
Laboratory data changes | 112 days
  Biochemistry, Hematology, Urinalysis
AE incidences over the study period | 112 days
  AE recording
Incidence of treatment related AE with ≥ Grade 2 | 112 days
  Incidence of subjects experiencing treatment related AE with ≥ Grade 2 according to the predefined toxicity grading scale in this study
Changes in physical examinations | 112 days
  Changes in physical examinations
Changes in vital signs | 112 days
  Changes in vital signs
Changes of ECG examination results | 112 days
  Changes of ECG examination results

CONTACTS AND LOCATIONS:
Overall Officials: Ken Hung, Ph.D., Study Director — Virginia Contract Research Organization Co., Ltd.
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No